CLINICAL TRIAL: NCT03739723
Title: The Surgical Education Culture Optimization Through Targeted Interventions Based on National Comparative Data (SECOND) Trial
Brief Title: The Surgical Education Culture Optimization Through Targeted Interventions Based on National Comparative Data - "The SECOND Trial"
Acronym: SECOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American College of Surgeons (Other); American Board of Surgery (Other); Accreditation Council for Graduate Medical Education (Other)
Responsible Party: Principal Investigator, Karl Bilimoria, MD, Professor of Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SECOND Trial
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Surgical Residency; Workplace Culture; Mistreatment; Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Programs will continue to conduct normal educational activities.
- Intervention Arm (Experimental): The intent of the intervention arm is to provide programs with data and resources to inform and improve surgical learning environments and resident wellness.
  Interventions: Other: Resource allocation to improve surgical learning environments

INTERVENTIONS:
Other: Resource allocation to improve surgical learning environments — If a hospital/program is assigned to the intervention arm, they will receive numerous resources including a program-specific learning environment and resident well-being report, a Wellness Toolkit, coaching webinars, and in-person/virtual conferences to help improve their surgery learning environment and residents' well-being.
  Arms: Intervention Arm

SUMMARY:
Due to a number of factors, residents are susceptible to mistreatment (i.e., discrimination, harassment, and abuse) and toxic outcomes (i.e., burnout, attrition, and suicidality). Our work following the FIRST Trial identified considerable variation in program-level rates of resident-reported burnout, gender discrimination, racial discrimination, sexual harassment, and verbal abuse. To investigate these issues, the SECOND Trial will include a national mixed-methods analysis of and a pragmatic cluster-randomized controlled trial to improve the resident learning environment and trainee wellness.

DETAILED DESCRIPTION:
The prospective, pragmatic cluster-randomized controlled trial will include approximately 320 surgical training programs across the United States. Participating programs will be randomized to the intervention or control arm. The intervention arm (vs. control) will receive program-specific reports about their learning environment and residents' well-being, as well as access to a Wellness Toolkit of ready-to-implement interventions. We will provide implementation support help facilitate and support intervention uptake throughout the trial period.

To assess the individual efficacy of the reports in regards to decreasing rates of mistreatment and toxic outcomes, the reports will be given to programs approximately 2 months to 6 months prior to Toolkit dissemination. Prior to Toolkit dissemination, programs will have the opportunity to fully review the report, form internal teams to address the issues, and mobilize necessary resources in preparation for receiving the Toolkit. A comprehensive list of all activities performed after report dissemination will be kept at a program-level. Toolkit dissemination to intervention programs will occur within 6 months of report dissemination. Coaching webinars and in-person/virtual conferences will be held at a variety of time points during the trial. The control arm will continue to perform their normal educational (including potential wellness) activities.

The investigators will compare multiple outcomes between the two study arms using data collected from an annual resident survey.

Extension of this work is anticipated to surgical subspecialty training programs (e.g., vascular surgery, cardiothoracic surgery). Eligible subspecialty programs will be assigned as per the randomization scheme of corresponding general surgery programs at their institution. Similar protocols will be in place for surgical subspecialties, with modifications to investigate specialty-specific survey items and interventions.

ELIGIBILITY:
Inclusion Criteria:

* Surgery training programs in the United States

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Burnout | 1 Year
  The primary outcome for the trial is reported rates of general surgery resident burnout.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Surgical Outcomes and Quality Improvement Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Janczewski LM, Buchheit JT, Golisch KB, Amortegui D, Mackiewicz N, Eng JS, Turner PL, Johnson JK, Bilimoria KY, Hu YY. Contemporary Evaluation of Work-Life Integration and Well-Being in US Surgical Residents: A National Mixed-Methods Study. J Am Coll Surg. 2024 Dec 1;239(6):515-526. doi: 10.1097/XCS.0000000000001135. Epub 2024 Nov 15. PMID 38920301
- See also: Flexibility In duty hour Requirements for Surgical Trainees Trial - "The FIRST Trial" — https://thefirsttrial.org/
- See also: Surgical Education Culture Optimization through targeted interventions based on National comparative Data (SECOND) Trial — http://thesecondtrial.org/

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT03739723/SAP_000.pdf